CLINICAL TRIAL: NCT07259681
Title: Intestinal Microbiome Profiles in Women With Gynecological Tumors and Pelvic Toxicity Secondary to Radiotherapy and Chemotherapy: Comparison With Controls and Effect of Rectal Ozone Treatment.
Brief Title: Gut Microbiome in Gynecological Cancer Patients With Pelvic Toxicity: Controls Versus Ozone Treatment. (MicrOzoGineTox)
Acronym: MicrOGineTox
Status: Not yet recruiting | Type: Observational
Sponsor: Bernardino Clavo, MD, PhD (Other)
Collaborators: Dr. Negrin University Hospital (Other); Complejo Hospitalario Universitario Insular Materno Infantil (CHUIMI) (Unknown); Fundacion Canaria Instituto de Investigacion Sanitaria de Canarias (Other); Instituto Universitario de Enfermedades Tropicales y Salud Pública de Canarias, Universidad de La Laguna (Unknown); CIBER (Infectious diseases) (Unknown)
Responsible Party: Sponsor-Investigator, Bernardino Clavo, MD, PhD, Principal Investigator, Research Unit Director, Dr. Negrin University Hospital
Organization: Dr. Negrin University Hospital (Other)
Other Study IDs: 2025-436-1; PIFIISC25/52 (Other Grant/Funding Number: FIISC (Fundación Canaria Inst. Investig. Sanitaria Canarias)); CIGC'25/26 (Other Grant/Funding Number: Cabildo de Gran Canaria (CIGC))
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-11

CONDITIONS: Pelvic Toxicity; Radiation Toxicity; Chemotherapy Toxicity; Gynecological Tumors; Radiation Proctitis; Radiation Cystitis; Vaginal Mucositis; Vulvar Mucositis; Quality of Life; Dysbiosis
Keywords: Gut microbiota; Ozone; Ozone therapy; Gynecological tumors; Radiotherapy; Chemotherapy; Side effects; Actinic proctitis; Actinic cystitis; Quality of life; Dysbiosis
MeSH Terms: conditions — Radiation Injuries; Dysbiosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Biospecimen Retention: Samples With DNA — Stool and serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TPIRQT Group (Cases): Patients with gynecological tumors treated with RT and/or CT who develop chronic pelvic toxicity (TPIRQT) and are referred for compassionate-use rectal ozone therapy at the Chronic Pain Unit. Samples and data will be collected before and after ozone therapy
- Control Group: pelvic toxicity (TPIRQT). This group will be matched by age (± 5 years) and primary tumor location. Samples and data will be collected once during a follow-up visit.

SUMMARY:
Patients treated for gynecological tumors with radiotherapy (RT) and/or chemotherapy (CT) frequently develop pelvic toxicity (TPIRQT), a condition that can become persistent, progressive, and refractory to standard treatments. This toxicity, affecting the rectum (proctitis), bladder (cystitis), and vagina (mucositis), severely deteriorates quality of life. Standard options for refractory cases are limited; at our center, rectal ozone therapy is used with high rates of symptomatic improvement (66-75%). Emerging evidence suggests a link between gut microbiota and the development of TPIRQT. However, it is unknown how rectal ozone therapy may influence the gut microbiome or if this modulation is part of its therapeutic mechanism. This prospective observational study will investigate the potential relationship between gut microbiome profiles (composition and diversity), the presence and severity of TPIRQT, and the response to rectal ozone therapy.

DETAILED DESCRIPTION:
Patients treated for gynecological tumors with radiotherapy (RT) and/or chemotherapy (CT) frequently develop pelvic toxicity (TPIRQT), a condition that can become persistent, progressive, and refractory to standard treatments. This toxicity, affecting the rectum (proctitis), bladder (cystitis), and vagina (mucositis), severely deteriorates quality of life. Standard options for refractory cases are limited; at our center, rectal ozone therapy is used with high rates of symptomatic improvement (66-75%). Emerging evidence suggests a link between gut microbiota and the development of TPIRQT. However, it is unknown how rectal ozone therapy may influence the gut microbiome or if this modulation is part of its therapeutic mechanism. This prospective observational study will investigate the potential relationship between gut microbiome profiles (composition and diversity), the presence and severity of TPIRQT, and the response to rectal ozone therapy.

ELIGIBILITY:
Inclusion Criteria for all patients (Cases and Controls):

1. Adult women (>=18 years).
2. Diagnosed with gynecological tumors (any location and stage).
3. Previously treated with radiotherapy and/or chemotherapy.
4. Must accept and sign the specific informed consent for this study.

   Additional Inclusion Criteria for inclusion in the TPIRQT Group (Cases):
5. Must present chronic TPIRQT with >= 3 months of duration after habitual symptomatic treatment.
6. Must have a toxicity Grade of 2 (moderate symptoms, limiting instrumental ADL) or higher, according to the CTCAE v.5.0 scale.

Exclusion Criteria for all patients (Cases and Controls):

1. Not meeting all inclusion criteria.
2. Presence of active inflammatory bowel disease (e.g., Crohn's Disease, Ulcerative Colitis) or a history of major gastrointestinal resection (excluding appendectomy) that could significantly alter gut anatomy and microbiota.
3. Any uncontrolled intercurrent illness or psychiatric condition that, in the investigator's opinion, would limit compliance with study requirements or interfere with the interpretation of results.
4. Unwillingness or inability to provide written informed consent for study participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with gynecological tumors treated with RT and/or CT with or without chronic pelvic toxicity (TPIRQT).
Sampling Method: Non-Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-01-15 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of gut microbiome profile (composition and diversity) between TPIRQT and Control groups | Baseline (single time point for controls, pre-ozone for cases)
  Gut microbiome composition and diversity (from a single sample) in control patients will be compared to the baseline profile of patients with TPIRQT.
Change in gut microbiome profile (composition and diversity) in patients with TPIRQT after rectal ozone therapy. | Baseline (pre-ozone therapy) , 4 Months (post-ozone therapy)
  Gut microbiome composition and diversity will be analyzed from stool samples using 16S ribosomal RNA gene sequencing.
Correlation of gut microbiome profile with grade of pelvic toxicity. | Baseline (for Control group); Baseline, 4 Months (for TPIRQT group).
  Toxicity will be assessed using: i) the CTCAE v.5.0 scale from the NCI , and ii) the EORTC QLQ-CX24 questionnaire. This will be evaluated for its relationship to microbiome data.

SECONDARY OUTCOMES:
Correlation of gut microbiome profile with health-related quality of life (HRQoL). | Baseline (for Control group); Baseline, 4 Months (for TPIRQT group).
  HRQoL will be assessed using: i) the EQ-5D-5L questionnaire, and ii) the EORTC QLQ-C30 questionnaire. This will be evaluated for its relationship to microbiome data.
Correlation of gut microbiome profile with anxiety and depression levels. | Baseline (for Control group); Baseline, 4 Months (for TPIRQT group).
  Anxiety and depression will be assessed using the Hospital Anxiety and Depression Scale (HADS). This will be evaluated for its relationship to microbiome data.
Correlation of gut microbiome profile with biochemical markers of oxidative stress and inflammation. | Baseline (for Control group); Baseline, 4 Months (for TPIRQT group).
  Serum samples will be collected to analyze biochemical parameters of oxidative stress and inflammation and their potential relationship with gut microbiome composition.

CONTACTS AND LOCATIONS:
Overall Officials: Bernardino Clavo, MD, PhD, Study Chair — Hospital Universitario de Gran Canaria Dr. Negrín, (FIISC), Las Palmas, Spain; Jacob Lorenzo-Morales, Prof, Principal Investigator — Instituto Universitario de Enfermedades Tropicales y Salud Publica de Canarias, Universidad La Laguna; Francisco Rodríguez-Esparragón, BSc, PhD, Principal Investigator — Hospital Universitario de Gran Canaria Dr. Negrín, (FIISC), Las Palmas, Spain
Locations (2):
- Spain (2):
  - Hospital Universitario de Gran Canaria Dr. Negrín, (FIISC), Las Palmas de Gran Canaria, Las Palmas
  - Instituto Universitario de Enfermedades Tropicales y Salud Pública de Canarias - Universidad de La Laguna, San Cristóbal de La Laguna, Tenerife

IPD SHARING:
Plan to Share IPD: Yes
* It will be available (after request): Individual participant data (IPD) that underlie the results reported in further articles, after deidentification
  * Data will be available after publication, ending 36 months following article publication.
  * They will be available for investigators whose proposed use of the data has been apd by an independent review committee identified for this purpose.
Time Frame: Data will be available after publication, ending 36 months following article publication.
Access Criteria: They will be available for investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose

REFERENCES:
- [Background] Clavo B, Canovas-Molina A, Ramallo-Farina Y, Federico M, Rodriguez-Abreu D, Galvan S, Ribeiro I, Marques da Silva SC, Navarro M, Gonzalez-Beltran D, Diaz-Garrido JA, Cazorla-Rivero S, Rodriguez-Esparragon F, Serrano-Aguilar P. Effects of Ozone Treatment on Health-Related Quality of Life and Toxicity Induced by Radiotherapy and Chemotherapy in Symptomatic Cancer Survivors. Int J Environ Res Public Health. 2023 Jan 13;20(2):1479. doi: 10.3390/ijerph20021479. PMID 36674232
- [Background] Clavo B, Navarro M, Federico M, Borrelli E, Jorge IJ, Ribeiro I, Rodriguez-Melcon JI, Carames MA, Santana-Rodriguez N, Rodriguez-Esparragon F. Long-Term Results with Adjuvant Ozone Therapy in the Management of Chronic Pelvic Pain Secondary to Cancer Treatment. Pain Med. 2021 Sep 8;22(9):2138-2141. doi: 10.1093/pm/pnaa459. No abstract available. PMID 33738491
- [Background] Clavo B, Navarro M, Federico M, Borrelli E, Jorge IJ, Ribeiro I, Rodriguez-Melcon JI, Carames MA, Santana-Rodriguez N, Rodriguez-Esparragon F. Ozone Therapy in Refractory Pelvic Pain Syndromes Secondary to Cancer Treatment: A New Approach Warranting Exploration. J Palliat Med. 2021 Jan;24(1):97-102. doi: 10.1089/jpm.2019.0597. Epub 2020 May 5. PMID 32379556
- [Background] Clavo B, Santana-Rodriguez N, Llontop P, Gutierrez D, Ceballos D, Mendez C, Rovira G, Suarez G, Rey-Baltar D, Garcia-Cabrera L, Martinez-Sanchez G, Fiuza D. Ozone Therapy in the Management of Persistent Radiation-Induced Rectal Bleeding in Prostate Cancer Patients. Evid Based Complement Alternat Med. 2015;2015:480369. doi: 10.1155/2015/480369. Epub 2015 Aug 18. PMID 26357522
- [Background] Clavo B, Ceballos D, Gutierrez D, Rovira G, Suarez G, Lopez L, Pinar B, Cabezon A, Morales V, Oliva E, Fiuza D, Santana-Rodriguez N. Long-term control of refractory hemorrhagic radiation proctitis with ozone therapy. J Pain Symptom Manage. 2013 Jul;46(1):106-12. doi: 10.1016/j.jpainsymman.2012.06.017. Epub 2012 Oct 26. PMID 23102757
- [Background] Wang A, Ling Z, Yang Z, Kiela PR, Wang T, Wang C, Cao L, Geng F, Shen M, Ran X, Su Y, Cheng T, Wang J. Gut microbial dysbiosis may predict diarrhea and fatigue in patients undergoing pelvic cancer radiotherapy: a pilot study. PLoS One. 2015 May 8;10(5):e0126312. doi: 10.1371/journal.pone.0126312. eCollection 2015. PMID 25955845
- [Background] Wang L, Wang X, Zhang G, Ma Y, Zhang Q, Li Z, Ran J, Hou X, Geng Y, Yang Z, Feng S, Li C, Zhao X. The impact of pelvic radiotherapy on the gut microbiome and its role in radiation-induced diarrhoea: a systematic review. Radiat Oncol. 2021 Sep 25;16(1):187. doi: 10.1186/s13014-021-01899-y. PMID 34563216
- [Background] Li L, Yang Z, Yi Y, Song Y, Zhang W. Gut microbiota and radiation-induced injury: mechanistic insights and microbial therapies. Gut Microbes. 2025 Dec;17(1):2528429. doi: 10.1080/19490976.2025.2528429. Epub 2025 Jul 6. PMID 40618373
- [Background] Ma CY, Zhao J, Xu XT, He XL, Qin SB, Zhou JY. Predictive biomarkers in the gut microbiome and metabolome for severe acute radiation enteritis in cervical cancer radiotherapy. Discov Oncol. 2025 Jul 1;16(1):1220. doi: 10.1007/s12672-025-03077-y. PMID 40591053